CLINICAL TRIAL: NCT06329427
Title: Dragon Ambient eXperience (DAX) Express Pilot Evaluation
Brief Title: Dragon Ambient eXperience (DAX) Copilot Evaluation
Acronym: DAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Hieu Nguyen, MS - Biostatician (Unknown); McKenzie Isreal, MPH - project manager (Unknown); Casey Stephens, MPH - Health services researcher (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00098063
Record Dates: First submitted 2024-03-18; First posted 2024-03-26 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Automated Clinical Documentation
Keywords: speech-to-text; Dragon Ambient eXperience (DAX); intervention evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Dragon Ambient eXperience (DAX) (Active Comparator): Clinicians interacted with DAX Copilot
  Interventions: Other: Dragon Ambient eXperience (DAX) Copilot
- No Intervention - Control group (No Intervention): Clinicians with standard care

INTERVENTIONS:
Other: Dragon Ambient eXperience (DAX) Copilot — The tool (DAX) listens to the conversation between a clinician and patient/caregiver during their visit, provides transcriptions between different speakers for the clinician to review, edit, and included in the final EHR notes.
  Other Names: Dragon Ambient eXperience (DAX)
  Arms: Intervention - Dragon Ambient eXperience (DAX)

SUMMARY:
AI solutions like, Dragon Ambient eXperience (DAX) Copilot (Nuance/Microsoft), hold the potential to significantly enhance provider and patient interactions and alleviate pain points that contribute to burn out. Atrium Health was the first healthcare system in the world to pilot Nuance's DAX Copilot intelligence (AI) enabled scribe software, which synthesizes a draft clinic note by "listening" to the conversation between a provider and patient. After 180 days of use by primary care clinicians and advanced practice providers (APPs), along with a control group, the investigators assess provider satisfaction, patient experience, and provider efficiency through qualitative and quantitative methods.

DETAILED DESCRIPTION:
In this non-randomized stepped-wedge trial, clinicians (including physicians and advanced practice providers [APP]) specializing in family medicine, internal medicine, and general pediatrics were recruited from outpatient clinics located in North Carolina and Georgia. The intervention group was divided into 5 waves between June and August 2023 based on clinic locations. Prior to the activation of accounts, clinicians underwent a one-hour training session on DAX Copilot. Meanwhile, a comparison group comprising clinicians not utilizing DAX was recruited in five waves from locations and specialties similar to those of the intervention group. Two types of primary outcomes, electronic health record (EHR) metrics and financial metrics, were assessed after 180 days of intervention. EHR metrics include time in EHR (EHR8), work time outside of work (WOW8), time in documentation (Note8), completed appointment rate, same day closure rate, and note length. Financial metrics include gross revenue per visit and work relative value units (wRVU) per visit. Secondary outcome include provider satisfaction survey, provider interview, and patient satisfaction survey.

ELIGIBILITY:
Inclusion Criteria:

* clinicians specializing in family medicine, internal medicine, and general pediatrics (including physicians and advanced practice providers [APPs])
* (intervention group) showed interests in participating in Dragon Ambient eXperience (DAX) Copilot
* (control group) clinicians who opted out from Dragon Ambient eXperience (DAX) Copilot in vendor's baseline survey
* (control group) clinicians who worked in the same clinic/region as the intervention group

Exclusion Criteria:

* preceptors
* inactive DAX participants (i.e., had DAX license but never activate it)
* have the same first use and last use DAX date
* missing demographics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Total EHR time | Month 10
  Total time on EHR (during and outside of clinic sessions) per 8 hour of patient scheduled time.
Work outside of work | Month 10
  Time on EHR outside of scheduled patient hours per 8 hour of patient scheduled time.
Time on encounter note documentation | Month 10
  Hours on documentation (note writing) per 8 hour of scheduled patient time
Completed appointment rate | Month 10
  Total completed visits over scheduled visits
Same day closure rate | Month 10
  Number of visits closed on the same day over total scheduled visits
Note length | Month 10
  Length of note in EPIC for each visit
Gross revenue per visit | Month 10
  Total charged amount in each day over total completed visits on the same day
wRVU per visit | Month 10
  Total work relative value units (wRVU) in each day over total completed visits on the same day

SECONDARY OUTCOMES:
Provider satisfaction | Month 4
  REDCap survey to clinicians in both groups (intervention and control) and assess their satisfaction of the new tool.
Provider interview | Month 1
  12 semi-structured interview on clinicians in the intervention group. Each interview was facilitated using an interview guide with a semi-structured list of questions to help guide the conversation and answer the learning objectives.
Patient satisfaction | Month 6
  Patient satisfaction on the visit - patient satisfaction surveys are collected as part of routine care, which will be accessed through Medallia. Scores range between 0 (worst) to 10 (best) with one decimal point.

CONTACTS AND LOCATIONS:
Overall Officials: Tsai-Ling Liu, PhD, Principal Investigator — Wake Forest University Health Sciences; Timothy C Hetherington, MS, Principal Investigator — Wake Forest University Health Sciences; Jeffrey A. Cleveland, MD, FAAP, Study Chair — Wake Forest University Health Sciences
Locations (5):
- United States (5):
  - Atrium Health Navicent, Macon, Georgia
  - Atrium Health Floyd, Rome, Georgia
  - Atrium Health, Charlotte, North Carolina
  - Scotland Health Care System, Laurinburg, North Carolina
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No